CLINICAL TRIAL: NCT00136214
Title: A Study of the Cerebral Effect of Pegylated Interferon in Hepatitis C Positive Subjects
Brief Title: Cerebral Effects of Pegylated Interferon in Hepatitis C Positive Subjects
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Schering-Plough (Industry)
Responsible Party: Principal Investigator, Nezam H. Afdhal, Professor of Medicine, Part-time, Beth Israel Deaconess Medical Center
Other Study IDs: 2003P000341
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Results first posted 2018-07-12 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-06

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Interferon Treated Group: Group treated with PEG-Interferon and ribavirin and undergoing MR brain and neuropsychiatric tests
  Interventions: Diagnostic Test: MR brain and neuropsychiatric tests
- Non-treated cohort control: Group undergoing MR brain and neuropsychiatric tests
  Interventions: Diagnostic Test: MR brain and neuropsychiatric tests

INTERVENTIONS:
Diagnostic Test: MR brain and neuropsychiatric tests

SUMMARY:
The hypothesis of this study is that pegylated interferon would cause cognitive deficits and mood changes in hepatitis C (HCV) positive subjects.

DETAILED DESCRIPTION:
Subjects with non-cirrhotic hepatitis C will have a magnetic resonance imaging (MRI)/magnetic resonance (MR) spectroscopy and neuropsychological testing prior to starting interferon. Subjects will have repeat testing following 12 weeks of interferon therapy and again at 12 weeks post interferon therapy.

MR spectroscopy (MRS) will measure the cerebral metabolites, NAA (N-acetyl aspartate), Cho (choline), MI (myoinositol) and Cr (creatine) at 3 distinct brain regions, i.e. basal ganglia and 2 locations within the frontal cortex.

Neuropsychological testing will include tests of the following cognitive domains: executive functioning, memory, language, motor skills and will also include questionnaires pertaining to quality of life (SF-36), mood (Beck's depression inventory) and a self-rating cognitive questionnaire (Conners' Adult Attention Deficit Hyperactivity Disorder Rating Scales [CAARS]).

Control subjects will include non-cirrhotic HCV subjects who are not taking interferon therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years old) of both sexes with chronic HCV infection (all genotypes).
* Subjects due to start treatment with pegylated interferon-alpha (IFN-a) for HCV eradication.
* Subjects with chronic hepatitis C who have elected not to be treated with pegylated-IFN-a
* Subjects with mild fibrosis on liver biopsy (stage 0-III/IV fibrosis)
* Subjects able to give informed consent.
* Subjects with controlled depression currently taking anti-depressant medication.

Exclusion Criteria:

* Subjects with cirrhosis on liver biopsy.
* Subjects with active alcohol or drug abuse.
* Subjects co-infected with human immunodeficiency virus (HIV).
* Subjects with structural brain abnormality, past history of cerebrovascular accident (CVA) or serious head trauma.
* Subjects with seizure disorder.
* Subjects with any contraindication to IFN therapy.
* Subjects with a poor command of the English language.
* Subjects with a contraindication to MRI, e.g. pacemaker, claustrophobia.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HCV positive patients Subjects with cirrhosis, active alcohol or drug abuse, co-infection with human immunodeficiency virus (HIV), structural brain abnormality, past history of cerebrovascular accident (CVA), serious head trauma, and seizure disorder were excluded. Other exclusions were contraindication to PIFN therapy, current psychiatric disorder or contraindications to MRI e.g., pacemaker and claustrophobia.
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2004-03; Primary Completion 2008-01 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nezam Afdhal, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Byrnes V, Miller A, Lowry D, Hill E, Weinstein C, Alsop D, Lenkinski R, Afdhal NH. Effects of anti-viral therapy and HCV clearance on cerebral metabolism and cognition. J Hepatol. 2012 Mar;56(3):549-56. doi: 10.1016/j.jhep.2011.09.015. Epub 2011 Oct 23. PMID 22027578

RESULTS

PARTICIPANT FLOW:
Groups:
- Interferon Treated Group: Group treated with PEG-Interferon and ribavirin and undergoing MR brain and neuropsychiatric tests
  MR brain and neuropsychiatric tests
- Non-treated Cohort Control: Group undergoing MR brain and neuropsychiatric tests
  MR brain and neuropsychiatric tests
Period: Overall Study
Arm/Group | Interferon Treated Group | Non-treated Cohort Control
Started | 15 | 7
Completed | 15 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Interferon Treated Group | Non-treated Cohort Control | Total
Number analyzed (Participants) | 15 | 7 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 7 | 22
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 11 | 5 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 13 | 6 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 7 | 22

OUTCOME MEASURES:

1. Primary Outcome: Ratios of Cerebral Metabolites Choline (CH), Myoinisitol (MI) and N-acety Aspartate (NAA)to Creatine (Cr) in 3 Brain Regions Including Basal Ganglia, Frontal Cortex and Left Dorsolateral Prefrontal Cortex
Description: Evaluation of changes in MR spectroscopy. reductions in ratio of Cho and MI reflect improvements in cerebral inflammation and improvement in cognition. Increases in the NAA ratio are suggestive of improvement in cognitive function.
Time Frame: 18 months overall with measures performed at baseline (T1), week 12 (T2) and 12 weeks after end of treatment (T3) with PEG-IFN for 48 weeks which is 60 weeks post baseline
Population: One patient dropped out secondary to claustrophobia and was unable to complete MR portion of study
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- Interferon Treated Group: Group treated with PEG-Interferon and ribavirin and undergoing MR brain and neuropsychiatric tests
  MR brain and neuropsychiatric tests Significant reductions in basal ganglia Cho/Cr (p = 0.03) and basal ganglia MI/Cr (p = 0.03) were observed in sustained virological responders (SVRs, n = 8), but not non-responders/ relapsers (NR/R, n = 6), indicative of reduced cerebral infection and/or immune activation in those who cleared virus. SVRs demonstrated significant improvements in verbal learning, memory, and visuo-spatial memory.
- Non-treated Cohort Control: Group undergoing MR brain and neuropsychiatric tests
  MR brain and neuropsychiatric tests
  A small but significant improvement in neurocognitive function secondary to the practice effect was seen in both HCV controls and HCV subjects during treatment.
Arm/Group | Interferon Treated Group | Non-treated Cohort Control
Number analyzed (Participants) | 14 | 7
ratio
  Basal Ganglia, T1, Cho/Cr | 0.42 (0.26) | 0.30 (0.04)
  Basal Ganglia,T2, Cho/Cr | 0.28 (0.05) | 0.28 (0.05)
  Basal Ganglia, T3, Cho/Cr | 0.34 (0.18) | NA (NA) — time point not done as per protocol
  Basal Ganglia, T1, MI/Cr | 0.78 (0.19) | 0.78 (0.19)
  Basal Ganglia T2. MI/C | 0.71 (0.11) | 0.72 (0.21)
  Basal Ganglia T3, MI/C | 0.75 (0.13) | NA (NA) — time point not done as per protocol
  Frontal Cortex T1, Cho/Cr | 0.29 (0.12) | 0.28 (0.03)
  Frontal Cortex T2, Cho/Cr | 0.26 (0.03) | 0.29 (0.08)
  Frontal Cortex T3, Cho/Cr | 0.29 (0.06) | NA (NA) — time point not done as per protocol
  Basal Ganglia T1, NAA/Cr | 1.26 (0.27) | 1.28 (0.54)
  Basal Ganglia T2, NAA/Cr | 1.25 (0.03) | 1.07 (0.13)
  Basal Ganglia T3, NAA/Cr | 1.09 (0.17) | NA (NA) — time point not done as per protocol
  Frontal Cortex T1,Mi/Cr | 0.68 (0.14) | 0.77 (0.23)
  Frontal Cortex T2, MI/Cr | 0.75 (0.32) | 1.19 (0.68)
  Frontal Cortex T3, MI/Cr | 0.71 (0.36) | NA (NA) — time point not done as per protocol
  Frontal Cortex T1, NAA/Cr | 1.73 (0.29) | 1.55 (0.49)
  Frontal Cortex T2, NAA/Cr | 1.74 (0.25) | 1.72 (0.67)
  Frontal Cortex T3, NAA/Cr | 1.75 (0.37) | NA (NA) — time point not done as per protocol
  DLPFC T1, Cho/Cr | 0.31 (0.14) | 0.27 (0.05)
  DLPFC T2, Cho/Cr | 0.25 (0.04) | 0.27 (0.06)
  DLPFC T3, Cho/Cr | 0.26 (0.04) | NA (NA) — time point not done as per protocol
  DLPFC T1, MI/Cr | 0.79 (0.19) | 0.78 (0.18)
  DLPFC T2, MI/Cr | 0.75 (0.22) | 0.86 (0.13)
  DLPFC T3/ MI/Cr | 0.93 (0.41) | NA (NA) — time point not done as per protocol
  DLPFC T1, NAA/Cr | 1.72 (0.43) | 1.61 (0.31)
  DLPFC T2, NAA/Cr | 1.65 (0.28) | 1.60 (0.29)
  DLFPC T3, NAA/Cr | 1.78 (0.28) | NA (NA) — time point not done as per protocol
Statistical Analysis 1: Comparison: Interferon Treated Group; Within group comparison of IFN group for metabolites in basal ganglia Comparison on MR spectroscopy of Cho/Cr at time points 1,2 and 3; Test type: Superiority; p = 0.08, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Interferon Treated Group; Within group comparison of IFN group for metabolites in basal ganglia Comparison on MR spectroscopy of Mi/Cr at time points 1,2 and 3; Test type: Superiority; p = 0.3, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Interferon Treated Group; Within group comparison of IFN group for metabolites in basal ganglia Comparison on MR spectroscopy of NAA/Cr at time points 1,2 and 3; Test type: Superiority; p = 0.9, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Interferon Treated Group; Within group comparison of IFN group for metabolites in frontal cortex. Comparison on MR spectroscopy of Cho/Cr at time points 1,2 and 3; Test type: Superiority; p = 0.7, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Interferon Treated Group; Within group comparison of IFN group for metabolites in frontal cortex. Comparison on MR spectroscopy of MI/Cr at time points 1,2 and 3; Test type: Superiority; p = 0.4, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Interferon Treated Group; Within group comparison of IFN group for metabolites in frontal cortex. Comparison on MR spectroscopy of NAA/Cr at time points 1,2 and 3; Test type: Superiority; p = 0.6, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Interferon Treated Group; Within group comparison of IFN group for metabolites in DLPFC. Comparison on MR spectroscopy of Cho/Cr at time points 1,2 and 3; Test type: Superiority; p = 0.3, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Interferon Treated Group; Within group comparison of IFN group for metabolites in DLPFC. Comparison on MR spectroscopy ofMI/Cr at time points 1,2 and 3; Test type: Superiority; p = 0.3, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: Interferon Treated Group; Within group comparison of IFN group for metabolites in DLPFC. Comparison on MR spectroscopy of NAA/Cr at time points 1,2 and 3; Test type: Superiority; p = 0.3, Wilcoxon (Mann-Whitney)
Statistical Analysis 10: Comparison: Non-treated Cohort Control; Within group comparison of control group for metabolites in Basal ganglia. Comparison on MR spectroscopy of Cho/Cr at time points 1 and 2; Test type: Superiority; p = 0.4, Wilcoxon (Mann-Whitney)
Statistical Analysis 11: Comparison: Non-treated Cohort Control; Within group comparison of control group for metabolites in Basal ganglia. Comparison on MR spectroscopy of MI/Cr at time points 1 and 2; Test type: Superiority; p = 0.9, Wilcoxon (Mann-Whitney)
Statistical Analysis 12: Comparison: Non-treated Cohort Control; Within group comparison of control group for metabolites in Basal ganglia. Comparison on MR spectroscopy of NAA/Cr at time points 1 and 2; Test type: Superiority; p = 0.6, Wilcoxon (Mann-Whitney)
Statistical Analysis 13: Comparison: Non-treated Cohort Control; Within group comparison of control group for metabolites in frontal cortex. Comparison on MR spectroscopy of Cho/Cr at time points 1 and 2; Test type: Superiority; p = 0.7, Wilcoxon (Mann-Whitney)
Statistical Analysis 14: Comparison: Non-treated Cohort Control; Within group comparison of control group for metabolites in frontal cortex. Comparison on MR spectroscopy of MI/Cr at time points 1 and 2; Test type: Superiority; p = 0.1, Wilcoxon (Mann-Whitney)
Statistical Analysis 15: Comparison: Non-treated Cohort Control; Within group comparison of control group for metabolites in frontal cortex. Comparison on MR spectroscopy of NAA/Cr at time points 1 and 2; Test type: Superiority; p = 0.6, Wilcoxon (Mann-Whitney)
Statistical Analysis 16: Comparison: Non-treated Cohort Control; Within group comparison of control group for metabolites in DLPFC. Comparison on MR spectroscopy of Cho/Cr at time points 1 and 2; Test type: Superiority; p = 0.5, Wilcoxon (Mann-Whitney)
Statistical Analysis 17: Comparison: Non-treated Cohort Control; Within group comparison of control group for metabolites in DLPFC. Comparison on MR spectroscopy of MI/Cr at time points 1 and 2; Test type: Superiority; p = 0.4, Wilcoxon (Mann-Whitney)
Statistical Analysis 18: Comparison: Non-treated Cohort Control; Within group comparison of control group for metabolites in DLPFC. Comparison on MR spectroscopy of NAA/Crat time points 1 and 2; Test type: Superiority; p = 0.9, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Neurocognitive Tests for Cerebral Function
Description: A battery of pen and paper neurocognitive tests where subject means are reported compared to the normative Z score. Data is reported at baseline (T1), week 12 on treatment (T2) and 12 weeks after treatment (week 60, T3). Improvements are increases in the test result compared to baseline as determined against the Z score. tests performed included Hopkins learning trials (HVLT), a measure of of verbal learning and memory and the Roy-Osterrieth Complex figure test (ROCF) which evaluates visio-spatal abilities, memory, planning and working memory. Improvements in the score (increases in value compared, either less negative or more positive to the Z score) shown in the table are reflective of improvements in these neurocognitive parameters.
Time Frame: 18 months overall with measures performed at baseline (T1), week 12 (T2) and 12 weeks after end of treatment (T3) with PEG-IFN for 48 weeks which is 60 weeks post baseline and only done in treated group and not controls
Measure: Mean (Standard Deviation); unit: Z-score
Groups:
- Interferon Treated Group: Group treated with PEG-Interferon and ribavirin and undergoing neuropsychiatric tests
- Non-treated Cohort Control: Group undergoing neuropsychiatric tests
Arm/Group | Interferon Treated Group | Non-treated Cohort Control
Number analyzed (Participants) | 15 | 7
Z-score
  HVLT, Verbal Learning Total, T1 | -1.43 (0.78) | -2.0 (1.01)
  HVLT, Verbal Learning Total, T2 | -0.78 (1.3) | -1.16 (0.79)
  HVLT, Verbal Learning Total, T3 | -0.7 (0.79) | NA (NA) — not performed at time point 3 as per protocol
  ROCF, T1 | 0.34 (0.49) | -1.0 (1.31)
  ROCF, T2 | 0.15 (0.77) | 0.05 (1.22)
  ROCF,T3 | 0.33 (0.52) | NA (NA) — not performed at time point 3 as per protocol
Statistical Analysis 1: Comparison: Interferon Treated Group vs Non-treated Cohort Control; Comparison between controls and IFN treated at time point 1 on change between scores for HVLT; Test type: Superiority; p > 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Interferon Treated Group vs Non-treated Cohort Control; Comparison between controls and IFN treated at time point 1 on change between scores for ROCF; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Interferon Treated Group vs Non-treated Cohort Control; Comparison between controls and IFN treated at time point 2 on change between scores for HVLT; Test type: Superiority; p > 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Interferon Treated Group vs Non-treated Cohort Control; Comparison between controls and IFN treated at time point 2 on change between scores for ROCF; Test type: Superiority; p > 0.05, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Interferon Treated Group | Non-treated Cohort Control
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/7
Serious Adverse Events (participants affected / at risk) | 1/15 | 0/7
Other Adverse Events (participants affected / at risk) | 0/15 | 0/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interferon Treated Group (N=15) | Non-treated Cohort Control (N=7)
Fatigue, fu like symptoms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Intolerant to interferon

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No